CLINICAL TRIAL: NCT06993038
Title: COMparison of Adenosine Versus Diltiazem FOR Supraventricular Tachycardia in the ED (COMFORT-ED) - Pilot Trial
Brief Title: Adenosine vs Diltiazem for Treatment of SVT in the ED
Acronym: COMFORT-ED
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Anne E. Zepeski (Other)
Responsible Party: Sponsor-Investigator, Anne E. Zepeski, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 202412202
Record Dates: First submitted 2025-04-03; First posted 2025-05-28 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Supraventricular Tachycardia (SVT)
Keywords: diltiazem; adenosine; emergency medicine
MeSH Terms: conditions — Tachycardia, Supraventricular | interventions — Adenosine; Diltiazem

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adenosine (Active Comparator)
  Interventions: Drug: adenosine
- Diltiazem (Active Comparator)
  Interventions: Drug: diltiazem

INTERVENTIONS:
Drug: adenosine — IV adenosine at standard doses for SVT (6 mg, 12 mg)
  Arms: Adenosine
Drug: diltiazem — IV diltiazem at standard doses for SVT (0.25 mg/kg)
  Arms: Diltiazem

SUMMARY:
This is a small, pilot study with a primary goal of assessing patient perceptions of two medication treatments for supraventricular tachycardia in adult patients treated in the Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18 years and older)
2. Diagnosis of acute, stable SVT in the emergency department

Exclusion Criteria:

1. Receipt of IV AV-nodal blocking agents prior to study enrollment (includes adenosine, non-dihydropyridine calcium channel blockers, beta-antagonists in pre-hospital and/or hospital setting).
2. Reported or confirmed personal history of Wolff-Parkinson-White (WPW) syndrome
3. History of heart failure with reduce ejection fraction (HFrEF) (LVEF</= 40%)
4. Severe bronchoconstrictive lung disease
5. Prior hypersensitivity to study medication
6. Previously enrolled in pilot study
7. Pregnant
8. Incarcerated

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility outcome | From enrollment to the end of ED encounter (up to 24 hours).
  Patients with stable SVT are identified in the ED (Threshold >90%)
Feasibility outcome | From enrollment to the end of ED encounter (up to 24 hours).
  Eligible participants who provide consent to participate (Threshold >50%)
Feasibility outcome | From enrollment to the end of ED encounter (up to 24 hours).
  Participants who complete all study procedures (Threshold >80%)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Zepeski, PharmD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
We have no plans to share individual participant data, pursuant to local IRB approval and policies.